CLINICAL TRIAL: NCT04941066
Title: Cognitive Process-based Real-time fMRI Neurofeedback in MDD and Rumination
Acronym: CNF-rumination
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laureate Institute for Brain Research, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 2021-002
Record Dates: First submitted 2021-06-10; First posted 2021-06-28 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Depression; Anxiety
Keywords: neurofeedback; real-time fMRI; rumination
MeSH Terms: conditions — Depression; Anxiety Disorders; Rumination Syndrome

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to a cognitive process-based real-time fMRI neurofeedback (CNF) or a sham condition.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active neurofeedback (Experimental): Receiving feedback signals from the rumination-related brain functional connectivity.
  Interventions: Behavioral: Active neurofeedback
- Sham neurofeedback (Sham Comparator): Receiving artificially generated feedback signals.
  Interventions: Behavioral: Sham neurofeedback

INTERVENTIONS:
Behavioral: Active neurofeedback — The session will be done on an individual basis. The active group will receive neurofeedback training from the rumination-related brain functional connectivity.
  Arms: Active neurofeedback
Behavioral: Sham neurofeedback — The session will be done on an individual basis. The sham group will receive neurofeedback training from an artificially generated random feedback signal.
  Arms: Sham neurofeedback

SUMMARY:
The purpose of this study is to assess the feasibility and efficacy of real-time fMRI neurofeedback for rumination.

DETAILED DESCRIPTION:
Neuroimaging MRI techniques for measuring brain structure, tissue composition, and Blood Oxygenation Level Dependent functional Magnetic Resonance imaging (BOLD fMRI) will be used to measure task-dependent and task-independent brain hemodynamic and electrophysiological changes in human subjects with major depressive disorders (MDD).

After being informed about the study and potential risks, all participants giving written informed consent will undergo one session of the cognitive process-based fMRI neurofeedback (CNF) targeting the rumination-related brain functional connectivity, and a one-week follow-up. Participants will be randomized in a double-blind manner (participant and investigator) in a 1:1 ratio to Active (receiving feedback from their own brain activity) or Sham (receiving artificially generated feedback).

ELIGIBILITY:
Inclusion Criteria:

* Good general health
* DSM-5 diagnosis of major depressive disorder (MDD)

Exclusion Criteria:

General Exclusion Criteria:

* Pregnancy

Medical Conditions:

* Moderate to severe traumatic brain injury (>30 min. loss of consciousness or >24 hours posttraumatic amnesia) or other neurocognitive disorder with evidence of neurological deficits.
* Presence of co-morbid medical conditions not limited to but including cardiovascular (e.g., history of acute coronary event, stroke) and neurological diseases (e.g., Parkinson's disease), as well as pain disorders.
* Presence of an uncontrolled medical condition that is deemed by the investigators to interfere with the proposed study procedures, or to put the study participant at undue risk.

Psychiatric Disorders:

* Current severe suicidal ideation or attempt within the past 12 months.
* Psychosis
* Bipolar disorder
* Substance abuse or dependence within the previous 6 months

Contraindications for MRI:

* Bodily implants of unsafe paramagnetic materials such as pace-makers and aneurysm clips.
* Claustrophobia that is severe enough to preclude MRI scanning.

Medications:

* Evidence of recreational drug use from a urine test.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Functional connectivity change between precuneus and right temporoparietal junction (rTPJ) | Through study completion (average: 2 weeks)
  Functional connectivity between precuneus and rTPJ will be calculated and evaluated using fMRI BOLD percent signal change.
Changes in Brooding subscale of Ruminative Responses Scale (RRS) scores | Through study completion (average: 2 weeks)
  The RRS Brooding subscale is a self-report scale to measure brooding ruminative responses. A higher score indicates higher brooding ruminative responses with a maximum score of 20 and a minimum score of 5.

SECONDARY OUTCOMES:
Changes in Depression subscale of Ruminative Responses Scale (RRS) scores | Through study completion (average: 2 weeks)
  The RRS Depression subscale is a self-report scale to measure depressive ruminative responses. A higher score indicates higher ruminative responses with a maximum score of 48 and a minimum score of 12.
Changes in Reflection subscale of Ruminative Responses Scale (RRS) scores | Through study completion (average: 2 weeks)
  The RRS Reflection subscale is a self-report scale to measure reflective ruminative responses. A higher score indicates higher ruminative responses with a maximum score of 20 and a minimum score of 5.
Changes in sum of Brooding and Depression subscales of Ruminative Responses Scale (RRS) scores | Through study completion (average: 2 weeks)
  The RRS Brooding and Depression subscales are a self-report scale to measure brooding and depressive ruminative responses. A higher score indicates higher ruminative responses with a maximum score of 68 and a minimum score of 17.
Changes in total score of Ruminative Responses Scale (RRS) scores | Through study completion (average: 2 weeks)
  The RRS is a self-report scale to measure ruminative responses. A higher score indicates higher ruminative responses with a maximum score of 88 and a minimum score of 22.

OTHER OUTCOMES:
Changes in Montgomery-Asberg Depression Rating Scale (MADRS) scores | Through study completion (average: 2 weeks)
  The MADRS is an interviewer-rated scale to measure the severity of depressive symptoms. A higher score indicates severer depression with a maximum score of 60 and a minimum score of 0.
Changes in Hamilton Anxiety Rating Scale (HAM-A) scores | Through study completion (average: 2 weeks)
  The HAMA is an interviewer-rated scale to measure the severity of anxiety symptoms. A higher score indicates severer anxiety with a maximum score of 56 and a minimum score of 0.
Changes in Patient Health Questionnaire (PHQ-9) scores | Through study completion (average: 2 weeks)
  The PHQ-9 is a self-report scale to measure depressive symptoms. A higher score indicates severer depressive symptoms with a maximum score of 27 and a minimum score of 0.
Changes in State-trait Anxiety Inventory (STAI) scores | Through study completion (average: 2 weeks)
  The STAI is a self-report scale to measure anxiety symptoms. The higher score indicates the higher anxiety with a maximum score of 80 and a minimum score of 20.
Changes in Metacognitions Questionnaire (MCQ-30) scores | Through study completion (average: 2 weeks)
  The MCQ-30 is a self-report scale to assess individual differences in five factors important in the metacognitive model of psychological disorders. The five subscales of the MCQ-30 are: cognitive confidence, positive beliefs about worry, cognitive self-consciousness, negative beliefs about uncontrollability of thoughts and danger, and beliefs about the need to control thoughts. The higher scores indicating higher levels of unhelpful metacognitions with a maximum total score of 120 and a minimum score of 30.
Changes in Thought Control Questionnaire (TCQ) scores | Through study completion (average: 2 weeks)
  The TCQ is a self-report scale to assess the effectiveness of strategies used for the control of unpleasant and unwanted thoughts. The TCQ measures five factors that correspond to different strategies for controlling unwanted thoughts: Distraction; Social Control; Worry; Punishment; and Re-appraisal. The higher scores indicating the effectiveness of strategies for controlling unwanted thoughts with a maximum total score of 120 and a minimum score of 30.
Changes in Rosenberg Self-Esteem Scale (RSE) scores | Through study completion (average: 2 weeks)
  The RSE is a self-report scale to assess global self-worth by measuring both positive and negative feelings about the self. A higher score indicates a higher self-esteem with a maximum score of 30 and a minimum score of 0.
Changes in Temporal Experience Of Pleasure Scale (TEPS) scores | Through study completion (average: 2 weeks)
  The TEPS is a self-report scale to assess pleasure experience. Anticipatory abstract pleasure reflected the pleasure experienced in anticipation of something more abstract or broad in nature. Consummatory abstract pleasure was related to consummation of emotional experience of something that is more abstract in nature. A lower score indicates a higher anhedonia propensity with a maximum total score of 120 and a minimum score of 25.
Changes in Emotion Regulation Questionnaire (ERQ) scores | Through study completion (average: 2 weeks)
  The ERQ is a self-report scale to assess how they regulate their emotions. The ERQ measures two emotion regulation strategies: Cognitive reappraisal and Expressive suppression. The higher indicates the greater the use of that particular emotion regulation strategy with a maximum total score of 70 and a minimum score of 10.
Changes in Positive And Negative Affect Schedule Extended (PANAS-X) scores | Through study completion (average: 2 weeks)
  The PANAS-X is a self-report scale to assess emotional states. The PANAS-X measures 11 specific affects: Fear, Sadness, Guilt, Hostility, Shyness, Fatigue, Surprise, Joviality, Self-Assurance, Attentiveness, and Serenity. Scores on Joviality could range from 8 to 40, with high scores indicating high happiness. Scores on Fear/Hostility/Guilt/Self-Assurance could range from 6 to 30, with high scores indicating high fear/hostility/guilt/self-assurance. Scores on Sadness could range from 5 to 25, with high scores indicating high happiness/sadness. Scores on Attentiveness/Shyness/Fatigue could range from 4 to 20, with high scores indicating high attentiveness/shyness/fatigue. Scores on Serenity/Surprise could range from 3 to 15, with high scores indicating high serenity/surprise.
Credibility Expectancy Questionnaire (CEQ) score | Through study completion (average: 2 weeks)
  The CEQ is the most widely used measure of treatment credibility and expectancy in psychotherapy research. The CEQ will be administered after the full introduction of the intervention rationale and principles and after the experience of the intervention. The items are rated on 9-point scales ranging from 1 (Not at all logical/useful/confident) to 9 (Very logical/useful/confident), with a total score possible range of 6 to 54. A higher score indicates higher treatment credibility and expectancy.
Post Neurofeedback Questionnaire score | Through study completion (average: 2 weeks)
  This is a study original questionnaire assessing the blindness and pleasantness. The blindness item is rated from 0 to 10, with a possible range of 0 to 10. The lower score indicates the confidence of the blindness. The pleasantness item is rated from 0 to 10 , with a possible range of 0 to 10. A higher score indicates the pleasantness of the intervention. The challenging/difficulties items are rated from 0 to 10, with a possible total range of 0 to 20. A higher score indicates the challenges/difficulties of the intervention. The two successful items are rated from 0 to 10, with a possible range of 0 to 20. A higher score indicates the subjective evaluation of the success of the intervention. The four mental strategies items are rated from 0 to 10, with a possible range of 0 to 40. A higher score indicates the mental strategies used in the intervention were helpful.

CONTACTS AND LOCATIONS:
Overall Officials: Salvador Guinjoan, MD, PhD, Principal Investigator — Laureate Institute for Brain Research
Locations (1):
- Laureate Institute for Brain Research, Tulsa, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No